CLINICAL TRIAL: NCT03591861
Title: Therapeutic Targeting of Sex Differences in Pediatric Brain Tumor Glycolysis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low accrual
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201806141
Record Dates: First submitted 2018-06-20; First posted 2018-07-19 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Pediatric Brain Tumor
MeSH Terms: interventions — Diet, Ketogenic; Carmustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Ketogenic Diet (Experimental): * Caregivers (and participating children) attend intro ketogenic diet class (4 - 30 min lectures)
  * Clinic visit with neurologist, nurse, and dietitian prior to hospital admission and then once every 3 months
  * Laboratory studies prior to hospital admission and then at each follow-up visit
  * Hospital admission (3-5 day) to start the ketogenic diet
  * Standard of care chemotherapy with BCNU for up to 2 years
  * Ketogenic diet can continue for up to 2 years
  Interventions: Procedure: Ketogenic diet; Drug: BCNU

INTERVENTIONS:
Procedure: Ketogenic diet — * Children under 2 years will immediately start on a full calorie classical 3:1 ketogenic diet. The 3:1 ratio indicates that the diet contains 3 g of fat for every 1 g of protein + carbohydrate, which results in about 87% of calories coming from fat.
  * Children 2 years or older will skip breakfast and lunch on the day of admission but start a full calorie 3:1 ketogenic diet at dinner.
Drug: BCNU — -Standard of care
  Other Names: Carmustine; BiCNU

SUMMARY:
The investigators will develop the concept of a sex-specific therapeutic intervention for gliomas that is based upon dietary carbohydrate restriction. The investigators will integrate metabolomics tools and FDG-PET imaging to validate the ketogenic diet on a sex-specific basis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a recurrent primary brain tumor with no curative therapy available.
* Measurable disease using pediatric Response Assessment in Neuro-Oncology Criteria (RANO) criteria.
* Life expectancy > 12 weeks
* Prior treatment with radiation alone, chemotherapy alone or combined radiation and chemotherapy is allowed.
* Patient is < 21 years of age
* Normal bone marrow and organ function as defined below:

  * Leukocytes ≥ 3,000/mcL
  * Absolute neutrophil count ≥ 1,500/mcl
  * Platelets ≥ 100,000/mcl
  * Total bilirubin ≤ 1.5 x IULN
  * AST(SGOT)/ALT(SGPT) ≤ 3.0 x IULN
  * Creatinine ≤ IULN OR creatinine clearance ≥ 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
  * Normal room air oxygenation must be documented. If room air oxygen saturation is less than 97%, a diffusion capacity of carbon monoxide (DLCO) of greater than 80%, must be demonstrated.
* Karnofsky or Lansky performance score of ≥ 60
* Patients of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a female patient become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Patient does not have any of the following conditions as they are contraindicated for ketogenic diet:

  * Primary and secondary carnitine deficiency
  * Carnitine palmitoyltransferase I or II deficiency
  * Carnitine translocase deficiency
  * Mitochondrial β-oxidation defects
  * Pyruvate carboxylase deficiency
  * Glycogen storage diseases
  * Ketolysis defects
  * Ketogenesis defects
  * Porphyria
  * Prolonged QT syndrome
  * Liver insufficiency
  * Renal insufficiency
  * Pancreatic insufficiency
  * Pulmonary insufficiency
  * Hyper insulinism
* Pregnant and/or breastfeeding. Female patients of childbearing potential must have a negative pregnancy test within 14 days of study entry.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of combining a ketogenic diet with chemotherapy in children with relapsed brain tumors as measured by the number of patients who can recruited with 3 years | Through completion of enrollment of all participants (estimated to be 3 years)
  * The study will be defined as being feasible if all 15 patients can be recruited within 3 years
  * Please note that feasibility of the study is dependent on both primary outcome measures
Feasibility of combining a ketogenic diet with chemotherapy in children with relapsed brain tumors as measured by if at least 80% of the patients comply with the intervention | Up to 2 years
  -The study will be defined as being feasible if at least 80% of the patients comply with the intervention as defined as achieving 80% of the targeted level of ketosis as assessed from laboratory measures and 80% of the planned BCNU doses
  --Please note that feasibility of the study is dependent on both primary outcome measures

SECONDARY OUTCOMES:
Tolerability of combining a ketogenic diet with chemotherapy in male children with relapsed brain tumors versus female children with relapsed brain tumors as measured by toxicity | Up to 2 years
  * All toxicities will be summarized by noting the count of participants who experience each toxicity
  * The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be utilized for all toxicity reporting.
Tumor response of male children with relapsed brain tumors to a ketogenic diet combined with chemotherapy versus female children with relapsed brain tumors as measured by progression-free survival (PFS) | Up to 10 years
  * PFS is defined as the duration of time from start of treatment to time of radiographic progression or death due to any cause, whichever occurs first.
  * Progression will be defined by the Response Assessment in Neuro-Oncology (RANO) working group guideline.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Cluster, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu